CLINICAL TRIAL: NCT00551655
Title: Impact of Drug Therapy and Co-Morbidities on the Development of Renal Impairment in HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: AIDS Arms Inc. (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: COL109413
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-10

CONDITIONS: Human Immunodeficiency Viruses; Kidney Failure; HIV Infections
Keywords: Human Immunodeficiency Viruses; Glomerular Filtration Rate; Tenofovir; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Renal Insufficiency; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tenofovir (TDF)-containing regimens may be associated with decreasing renal function in HIV-infected patients concurrently treated with boosted PI's and/or have co-morbid conditions including diabetes mellitus, hypertension, anemia, hepatitis B, and hepatitis C.

DETAILED DESCRIPTION:
COL109413 is a Phase IV retrospective database study involving the review of medical records of approximately 850 HIV-infected patients treated at a single center (Peabody Health Clinic, Dallas, Texas) and followed for up to a 4-year period (2003-2006). Patients whose GFR decreased >25% from baseline (BL) will be identified and their disease and treatment characteristics will be compared to those of patients whose GFR did not change. GFR will be calculated by both the MDRD and the Cockcroft-Gault methods.

The following information will be noted: patient age, weight, gender, race/ethnicity, viral load, CD4 cell count, serum creatinine and other available laboratory data, start of HAART therapy (TDF - vs non-TDF-containing), changes in drug treatment, co-morbidities (hypertension, diabetes mellitus, anemia, hepatitis C virus or hepatitis B virus infection), drug treatment for co-morbidities and non-HIV-related illnesses, and adherence by prescription refill. The study endpoints will be: time from treatment initiation-to-event (GFR decrease >25% from BL) analysis between TDF-containing vs non-TDF-containing antiretroviral therapy; number of patients who convert from National Kidney Foundation-defined mild to moderate renal impairment or from moderate to severe renal impairment in the TDF vs non-TDF-treated patients; effect of co-morbidities and concomitant medications on time to GFR decrease >25% from BL.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients seen between 2003 and 2006

Exclusion Criteria:

* Fewer than two laboratory results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2007-05; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Rawlings, MD, Principal Investigator — AIDS Arms Inc.
Locations (1):
- Peabody Health Center, Dallas, Texas, United States

REFERENCES:
- [Background] Roling J, Schmid H, Fischereder M, Draenert R, Goebel FD. HIV-associated renal diseases and highly active antiretroviral therapy-induced nephropathy. Clin Infect Dis. 2006 May 15;42(10):1488-95. doi: 10.1086/503566. Epub 2006 Apr 11. PMID 16619164
- [Background] Izzedine H, Launay-Vacher V, Deray G. Antiviral drug-induced nephrotoxicity. Am J Kidney Dis. 2005 May;45(5):804-17. doi: 10.1053/j.ajkd.2005.02.010. PMID 15861345
- [Background] Ross MJ, Klotman PE. HIV-associated nephropathy. AIDS. 2004 May 21;18(8):1089-99. doi: 10.1097/00002030-200405210-00002. No abstract available. PMID 15166524
- [Background] Guo X, Nzerue C. How to prevent, recognize, and treat drug-induced nephrotoxicity. Cleve Clin J Med. 2002 Apr;69(4):289-90, 293-4, 296-7 passim. doi: 10.3949/ccjm.69.4.289. PMID 11996200
- [Background] Iglesias JI, Nasr SH, Markowitz GS, D'Agati VD. AIDS, nephrotic-range proteinuria, and renal failure. Kidney Int. 2006 Jun;69(11):2107-10. doi: 10.1038/sj.ki.5000408. No abstract available. PMID 16641932
- [Background] Coca S, Perazella MA. Rapid communication: acute renal failure associated with tenofovir: evidence of drug-induced nephrotoxicity. Am J Med Sci. 2002 Dec;324(6):342-4. doi: 10.1097/00000441-200212000-00011. PMID 12495304
- [Background] Antoniou T, Raboud J, Chirhin S, Yoong D, Govan V, Gough K, Rachlis A, Loutfy M. Incidence of and risk factors for tenofovir-induced nephrotoxicity: a retrospective cohort study. HIV Med. 2005 Jul;6(4):284-90. doi: 10.1111/j.1468-1293.2005.00308.x. PMID 16011534
- [Background] Schaaf B, Aries SP, Kramme E, Steinhoff J, Dalhoff K. Acute renal failure associated with tenofovir treatment in a patient with acquired immunodeficiency syndrome. Clin Infect Dis. 2003 Aug 1;37(3):e41-3. doi: 10.1086/376643. Epub 2003 Jul 22. PMID 12884188
- [Background] Karras A, Lafaurie M, Furco A, Bourgarit A, Droz D, Sereni D, Legendre C, Martinez F, Molina JM. Tenofovir-related nephrotoxicity in human immunodeficiency virus-infected patients: three cases of renal failure, Fanconi syndrome, and nephrogenic diabetes insipidus. Clin Infect Dis. 2003 Apr 15;36(8):1070-3. doi: 10.1086/368314. Epub 2003 Apr 4. PMID 12684922
- [Background] Creput C, Gonzalez-Canali G, Hill G, Piketty C, Kazatchkine M, Nochy D. Renal lesions in HIV-1-positive patient treated with tenofovir. AIDS. 2003 Apr 11;17(6):935-7. doi: 10.1097/00002030-200304110-00026. No abstract available. PMID 12660548
- [Background] Verhelst D, Monge M, Meynard JL, Fouqueray B, Mougenot B, Girard PM, Ronco P, Rossert J. Fanconi syndrome and renal failure induced by tenofovir: a first case report. Am J Kidney Dis. 2002 Dec;40(6):1331-3. doi: 10.1053/ajkd.2002.36924. PMID 12460055
- [Background] Levey AS, Coresh J, Balk E, Kausz AT, Levin A, Steffes MW, Hogg RJ, Perrone RD, Lau J, Eknoyan G; National Kidney Foundation. National Kidney Foundation practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Ann Intern Med. 2003 Jul 15;139(2):137-47. doi: 10.7326/0003-4819-139-2-200307150-00013. PMID 12859163
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Sokoll LJ, Russell RM, Sadowski JA, Morrow FD. Establishment of creatinine clearance reference values for older women. Clin Chem. 1994 Dec;40(12):2276-81. PMID 7988015
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613